CLINICAL TRIAL: NCT02277457
Title: Personalized Adaptive Radiation Therapy With Individualized Systemic Targeted Therapy (PARTIST) for Locally Advanced, Non-small Cell Lung Cancer With Genomic Driver Mutations
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Augusta University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2014.117; HUM00094166 (Other: University of Michigan)
Record Dates: First submitted 2014-10-24; First posted 2014-10-29 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-06

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Crizotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EGFR Mutation (Experimental): Patients with an identified EGFR mutation will receive PET (Positron Emission Tomography) - Adaptive RT (Radiation Therapy) plus concurrent Erlotinib followed by 1 year total of Erlotinib Treatment.
  Interventions: Radiation: PET-Adaptive RT; Drug: Erlotinib
- ALK Rearrangement (Experimental): Patients with an identified EGFR mutation will receive PET (Positron Emission Tomography) - Adaptive RT (Radiation Therapy) plus concurrent Crizotinib followed by 1 year total ofCrizotinib Treatment.
  Interventions: Radiation: PET-Adaptive RT; Drug: Crizotinib

INTERVENTIONS:
Radiation: PET-Adaptive RT — All patients will be treated with response-driven PET-adaptive RT. The radiation dose will be delivered in greater than or equal to 2.2 Gy per daily fraction to FDG-PET/CT-guided target volumes with the treatment duration limited to 30 fractions and total radiation dose limited to 66-80.4 Gy.
Drug: Erlotinib — 150 mg once daily
  Arms: EGFR Mutation
Drug: Crizotinib — 250 mg twice daily
  Arms: ALK Rearrangement

SUMMARY:
Hypotheses:

Short-term - Targeted therapy with erlotinib or crizotinib plus PART (Personalized Adaptive Radiation Therapy) will be safe and will yield favorable outcomes in patients with stage III, EGFR (Epidermal Growth Factor Receptor) + or ALK (Anaplastic Lymphoma Kinase) + NSCLC (Non-Small Cell Lung Cancer).

Long-term - In patients with stage III NSCLC harboring driver mutations, treatment with relevant targeted agents plus PART will improve both local-regional and systemic tumor control resulting in improved survival relative to standard chemoradiotherapy.

DETAILED DESCRIPTION:
The proposed trial is a pilot study that will accrue 30 patients with inoperable stage IIIA/B NSCLC harboring either an EGFR mutation (n=20) or an ALK rearrangement (n=10). Patients with EGFR+ tumors will be treated with erlotinib 150 mg orally QD; patients with ALK+ tumors will be treated with crizotinib 250 mg orally BID. Treatment consists of six weeks of concurrent PART plus erlotinib or crizotinib, followed by erlotinib or crizotinib for a total of 1 year. All patients will be treated with response-driven PART with dose intensified to the active (FDG-avid) region based on a mid-treatment FDG-PET/CT scan while maintaining dose limits for organs-at-risk. The primary endpoints will be PFS and OS. Primary analyses will be performed separately for ALK+ and EGFR+ patients. The secondary endpoint of treatment-related toxicity will focus on pneumonitis and esophagitis with a strict stopping rule in place.

Current standard therapy affords suboptimal outcomes for patients with locally advanced NSCLC due to both locoregional and distant recurrences. Since targeted therapy is more effective than chemotherapy in patients with relevant driver mutations, the best way to significantly improve outcomes in this subgroup of patients is to optimize systemic therapy with targeted agents while improving local control with PET-adapted, high-dose RT.

ELIGIBILITY:
Inclusion Criteria:

* Patients with FDG-avid (radioactive glucose) and pathologically proven stage IIA-IIB or IIIA-IIIB non-small cell lung cancer (according to AJCC [American Joint Committee on Cancer] staging, 7th edition).
* Patients with tumors that harbor either EGFR sensitizing mutations or ALK rearrangement.
* Patients must be considered unresectable or medically inoperable; patients who decline surgery are also eligible.
* Patients must be 18 years of age or older.
* Patients with ECOG (Eastern Cooperative Oncology Group) performance status of 0-2.
* Patients must have adequate organ function.
* Patients must be able to take oral medications.
* Women with reproductive capability must be willing to use effective contraception.
* Patients must be informed of the investigational nature of this study and sign written informed consent in accordance with institutional and federal guidelines.
* Patients must be willing to comply with study procedures.

Exclusion Criteria:

* Patients with tumors that have a component of small cell carcinoma.
* Patients wtih stage I, II, or IV disease, including malignant pleural or pericardial effusion.
* Prior radiotherapy to the thorax such that composite radiation would significantly over-dose critical structures, either per estimation of the treating radiation oncologist or defined by failure to meet normal tissue tolerance constraints.
* Patients who cannot tolerate thoracic radiotherapy or targeted therapy.
* Patients wtih a prior diagnosis of interstitial lung disease or pulmonary fibrosis.
* Patients who cannot take oral medication, require intravenous alimentation, had prior surgical procedures affecting gastrointestinal absorption, or have active peptic ulcer disease.
* Hypersensitivity to erlotinib, crizotinib, or to any of the excipients.
* Pregnant women are excluded from this study because radiation has the potential for teratogenic or abortifacient effects.
* Prisoners are excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09; Primary Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Time to Progression From the Initiation of Study Treatment For ALK + and EGFR + Patients | 5 Years
Time to Death From Initiation of Study Treatment For ALK + and EGFR + Patients | 5 Years

SECONDARY OUTCOMES:
The Number of Patients Experiencing Pneumonitis and Esophagitis | 5 Years
The Number of Patients Experiencing Grade 3 or Higher Toxicities | 5 Years

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Kalemkerian, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States